CLINICAL TRIAL: NCT06288854
Title: Efficacy of Olanzapine on Weight Gain in Women with Advanced Stage Gynecologic Cancer Receiving Paclitaxel and Carboplatin Combination Chemotherapy : a Double Blind, Placebo-controlled Randomized Trial
Brief Title: Efficacy of Olanzapine on Weight Gain in Advanced Gynecologic Cancer with Paclitaxel and Carboplatin: a Double Blind, Placebo-controlled Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 66222
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-03

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: olanzapine vs placebo
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine (Experimental): Olanzapine 5 mg oral OD
  Interventions: Other: weight gain each group
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: weight gain each group

INTERVENTIONS:
Other: weight gain each group — weight gain after 12 Weeks
  Other Names: body weight

SUMMARY:
* Efficacy of olanzapine on weight gain in advanced stage gynecologic cancer
* Proprotion of pateints in advanced stage gynecologic cancer who recieving paclitaxel and carboplatin chemotherapy gain weight on olanzapine or placebo

DETAILED DESCRIPTION:
-Proprotion of pateints in advanced stage gynecologic cancer who recieving paclitaxel and carboplatin chemotherapy gain weight on olanzapine or placebo

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage gynecologic cancer receiving Paclitaxel and carboplatin chemotherapy
* ECOG 0-1
* Normal CBC,Liver, renal function
* Communication in Thai language or Thai caregiver
* Inform consent

Exclusion Criteria:

* Pregnancy
* Active infection
* Bowel obstruction or history of bowel surgery
* On dopamine receptor antagonists or psychiatric or anticonvulsant medication
* Olanzapine allery
* Abnormal function of liver and renal
* Diabetic melitus or morbid obesity
* patient can't selfcare

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of olanzapine on weight gain in advanzed stage gynecologic cancer recieving paclitexal and carboplatin chemotherapy | 12 weeks after intervention
  proprotion of pateints gain weight after intervention (olanzapine or placebo) by monitor weight before and after get intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code